CLINICAL TRIAL: NCT01544608
Title: A Non- Interventional Study to Observe Real Life Usage of Atypical Antipsychotics in the Acute Inpatient Management of Schizophrenia.
Brief Title: Observe Real-life Allocation of Atypical Antipsychotics in the Acute Inpatient Management of Schizophrenia
Acronym: RECONNECT-S
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-NME-XXX-2011/1
Record Dates: First submitted 2012-02-20; First posted 2012-03-06 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Acute psychotic episode of Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Subjects who are hospitalized due to acute psychotic episode.: All subjects who are hospitalized due to acute psychotic episode. The subjects should be managed according to normal clinical practice until discharge time.

SUMMARY:
The primary objective of this Non- Interventional Study (NIS) is to describe the use of atypical antipsychotics in subjects with Schizophrenia during the hospitalisation due to acute psychotic episode by evaluation of drug, dose and mode of administration of the medication.

DETAILED DESCRIPTION:
RECONNECT-S BETA

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for schizophrenia stated in The Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria.
* Subject is hospitalised due to an acute psychotic episode.
* Ability of the subject to understand and comply with the requirements of the study, as judged by the investigator.

Exclusion Criteria:

* Current participation in any clinical trial.
* Previous enrolment in the present NIS (in case of recurrence occurred during the enrolment period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric Institutes
Sampling Method: Non-Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Use of atypical antipsychotic(s) during hospitalisation. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.
Daily dosage of atypical antipsychotic(s) during hospitalisation. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.
Mode of administration of atypical antipsychotic(s) during hospitalisation. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.

SECONDARY OUTCOMES:
Percent of patients with atypical antipsychotic as monotherapy. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.
Percent of patients with combinations of antipsychotics. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.
Main criteria of an antipsychotic's selection during hospitalisation expressed as percentage. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.
Use of psychometric scales in day to day practice in therm of evaluation of the disease symptoms and thus efficacy of the treatment. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.
Description of the usage of concomitant psychiatric medication (other than atypical antipsychotic) during the hospitalization. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.
Relationship between medication used during the hospitalization and maintenance therapy recommended upon discharge. | Hospitalisation period, an expected average of 3 weeks (variable per patient).
  The data will be collected at one visit at the moment of discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Talaat Matar, CONSULTANT PSYCHIATRIST, Study Chair — Obaid Alla Hospital,Ras Al Khaima,UAE; Tarek Darwish, CONSULTANT PSYCHIATRIST, Study Chair — Sheikh Khalifa Medical City(SKMC), Abudhabi,UAE; Sohail Khan, CONSULTANT PSYCHIATRIST, Study Chair — Jeddah Psychiatric hospital,Jeddah, Saudi Arabia; Tarek Okasha, PROFESSOR, Study Chair — Ain Shams University, Cairo, Egypt; Mohamed Nasr, PROFESSOR, Study Chair — Cairo University, Egypt
Locations (7):
- Research Site, Cairo, Egypt
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- United Arab Emirates (3):
  - Research Site, Abu Dhabi
  - Research Site, Dubai
  - Research Site, Ras al-Khaimah